CLINICAL TRIAL: NCT06311539
Title: The Effect of Chronotype and Circadian Rhythm on Physical Performance in Healthy Male Individuals
Brief Title: The Effect of Circadian Rhythm on Physical Performance in Healthy Male Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Furkan Çakır, Principal Investigator, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IstanbulBUFC4
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Chronotype; Exercise
Keywords: circadian rhythm; chronotype; physical performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Outcomes Assessor
Masking Description: The evaluator who will perform isokinetic assessments and vertical jump measurements will be blinded to the participants' chronotype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning chronotype (Experimental): Participants who score between 59-70 in the Morningness Eveningness Questionnaire will be assigned to the morning chronotype group.
  Interventions: Other: Theraband Strengthening Exercise Program
- Evening chronotype (Experimental): Participants who score between 16-41 in the Morningness Eveningness Questionnaire will be assigned to the evening chronotype group.
  Interventions: Other: Theraband Strengthening Exercise Program

INTERVENTIONS:
Other: Theraband Strengthening Exercise Program — Resisted knee flexion in prone position and resisted knee extension in seated position (for dominant leg) and bilateral squats were practiced in 3 sets of 12 repetitions. Participants rested for 30 seconds between sets. The program, which lasted approximately 30 minutes in total, continued for a total of 6 weeks, the first 3 weeks with the red theraband and the last 3 weeks with the black theraband.
  15 morning type participants will be included in the morning exercise program (08:00) and 15 morning type participants will be included in the evening exercise program (18:00).
  15 evening type participants will be included in the morning exercise program (08:00) and 15 evening type participants will be included in the evening exercise program (18:00).

SUMMARY:
Little is known about optimizing the timing of exercise periods to maximize the health benefits of exercise. Furthermore, exercise is a potent modulator of skeletal muscle metabolism and it is clear that skeletal muscle has a robust circadian profile. Circadian rhythms can be observed in behavior, physiology, and metabolism. Various studies show that exercise changes the rhythm of the clock machines in skeletal muscle. Studies examining the relationship between exercise, especially strength training, and circadian rhythm are quite limited in the literature. Although some studies have shown that force peaks in the afternoon/evening hours, regardless of muscle group and contraction speed, there are no studies on how much this time interval varies from person to person and chronotype.

The aim of this study is to investigate to what extent strength training given at appropriate times for morning, evening and intermediate chronotypes creates changes in performance in healthy adult male individuals.

DETAILED DESCRIPTION:
After participants are informed about the research, evaluation and exercise protocol, their signed consent will be obtained.

The Morningness-Eveningness Questionnaire will be applied until 30 participants with morning type and 30 evening type chronotypes are reached. (Estimated for 100 students) After determining 30 morning type and 30 evening type participants, isokinetic evaluations will be made and vertical jump heights will be measured (T0).

Then, 15 morning type participants will be included in the morning exercise program (08:00) and 15 morning type participants will be included in the evening exercise program (18:00).

15 evening type participants will be included in the morning exercise program (08:00) and 15 evening type participants will be included in the evening exercise program (18:00).

Thus, some of the participants from both morning and evening groups will be included in strength training for 6 weeks, at a time appropriate to their chronotypes, and some at a time incompatible with their chronotypes. Isokinetic evaluations and vertical jump height measurements will be repeated at the end of the strengthening exercise program, which will last 3 days a week for 6 weeks, a total of 18 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Being male,
* Between the ages of 18-30
* Having a chronotype that was morning person or evening person in the Morningness-Eveningness Questionnaire

Exclusion Criteria:

* Being female
* Having an intermediate chronotype in the Morningness-Eveningness Questionnaire
* Having a history of surgery or limitation in the knee area
* Having a metabolic, neurological, or orthopedic disorder.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male participants will be included in the research.
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Isokinetic strength test | T0 and T1 (Baseline and after 6 week exercise program)
  Isokinetic evaluations will be made with the 'Biodex® System3 Isokinetic (Biodex Medical Systems, Inc, New York, New York, USA)' brand isokinetic dynamometer. The study will be performed on the dominant side lower extremity knee flexor and extensor muscle groups. Individuals' isokinetic quadriceps and hamstring muscle strengths will be evaluated at different angular velocities (60°/sec and 180°/sec). Quadriceps and hamstring muscle strengths will be evaluated with a protocol consisting of 5 repetitions of 60°/sec flexion-extension concentric-concentric movement, and 1 set of 10 repetitions of 180°/sec flexion-extension concentric-concentric movement. There will be 1-minute rest breaks between sets. Maximum voluntary contraction, peak torque and peak torque/body weight values will be recorded.
Vertical jump test | T0 and T1 (Baseline and after 6 week exercise program)
  For vertical jump height measurement, participants were asked to stand next to the wall on the dominant foot to be evaluated (jumping leg). The participant touched the wall, which was graded in centimeters, with one hand. The participant was asked to jump with all his strength and touch the highest point he could touch. The height of the jump made by the participant with the dominant foot was measured by recording the height of the vertical tip of the hand in the starting position and the test height. This test was repeated three times, with a 60-second rest interval between each jump. The best value obtained was recorded in centimeters (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Ilksan Demirbuken, PhD, Study Director — Marmara University, Faculty of Health Sciences; Ender Ersin Avci, PhD, Study Director — Marmara University, Faculty of Health Sciences; Mine Gulden Polat, PhD, Study Director — Marmara University

IPD SHARING:
Plan to Share IPD: No